CLINICAL TRIAL: NCT05026528
Title: Randomized Controlled Trial of a Digital Diabetes Self Management Education and Support System for Patients With Type 2 Diabetes in Primary Health Care
Brief Title: Digital Diabetes Self Management Education and Support for Patients With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis of primary outcome (HbA1c at 6 months) revealed no numerical differences after 80 included participants. Further inclusion of participants to reach prespecified N to evaluate primary outcome deemed futile. 138 participants included.
Sponsor: Region Jönköping County (Other Government)
Collaborators: Linkoeping University (Other Government); Region Östergötland (Other); Uppsala County Council, Sweden (Other Government); The Swedish Diabetes Foundation (Unknown); Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bra liv med diabetes typ 2
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: mHealth; Primary health care; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: An interim analysis comparing the change in HbA1c from baseline to six months between the two intervention groups was performed in march 2024 including 80 participants. The analysis was done according to intention-to-treat.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital DSME/S (Experimental): Ten-week intervention during which the participant uses a digital diabetes self management education and support system together with the diabetes nurse.
  Interventions: Other: Digital diabetes self management education and support system
- Standard care (No Intervention): Control group continuing with regular standardized care.

INTERVENTIONS:
Other: Digital diabetes self management education and support system — Digital diabetes self management and support system
  Other Names: Live well with type 2 diabetes
  Arms: Digital DSME/S

SUMMARY:
The purpose of this study is to test the effect of using a digital diabetes self management education and support system compared with standard care for patients with type 2 diabetes in primary health care.

DETAILED DESCRIPTION:
After being informed verbally and in text participants will sign a consent to participate. The participant will then be randomized to either use a digital diabetes self management education and support system for 10 weeks together with a diabetes nurse, or to continue with the regular care. The effects will be evaluated after 6, 12 and 36 months from randomization with emphasis on cardiovascular risk factors, life-style, diabetes knowledge and health economics.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus diagnosed according to WHO criteria < 5 years from randomization:
* Fasting plasma glucose > 7 mmol/L at two timepoints. OR
* HbA1c ≥ 48 mmol/mol twice or in combination with fasting plasma glucose > 7 mmo/L once. OR
* Non-fasting plasma glucose ≥ 11.1 mmol/L at one timepoint in combination with symptoms of hyperglycemia.
* Access to a digital ID-card to access the digital system
* Access to a computer, tablet or smart phone
* Sufficient knowledge of written and spoken Swedish to understand the information given in the digital system.

Exclusion Criteria:

* Treatment with Insulin
* Other co-morbidities limiting the use of the digital system according to the diabetes nurse judgement. E.g. dementia or severe psychiatric disease.
* Other forms of diabetes mellitus than type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  The level of glycated hemoglobin A1 in blood measured in mmol/mol.

OTHER OUTCOMES:
Plasma cholesterol | 6, 12 and 36 months
  mmol/L
Plasma LDL-cholesterol | 6, 12 and 36 months
  mmol/L
Plasma HDL-cholesterol | 6, 12 and 36 months
  mmol/L
Fasting plasma triglycerides | 6, 12 and 36 months
  mmol/L
Fasting plasma glucose | 6, 12 and 36 months
  mmol/L
Urinary albumin/creatinine ratio | 6, 12 and 36 months
  mg/mmol
Waist circumference | 6 and 12 months
  cm
Body mass index | 6, 12 and 36 months
  kg/m2
Self reported physical activity level | 6 and 12 months
  International Physical Activity Questionnaire (IPAQ)
Objectively measured physical activity level | 6 and 12 months
  Accelerometer Axivity AX3 will be used on a subgroup of 100 participants.
Self reported dietary intake | 6 and 12 months
  Indicator questions from the Swedish National Board of Health and Welfare
Health literacy | 6 and 12 months
  HLS-EU-Q16 questionnaire. 0-12 points. Higher score is better.
Patient-reported outcome and experience measures | 6 and 12 months
  Questionnaire developed and validated by the National Swedish Diabetes Registry. 0-100 points for each of 8 PROM scales and 4 PREM scales. Higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Stomby, MD/PhD, Principal Investigator — Region Jönköping County and Linköping University
Locations (15):
- Sweden (15):
  - Boxholms vårdcentral, Boxholm
  - Eksjö vårdcentral, Eksjö
  - Gislaved vårdcentral, Gislaved
  - Rosenhälsans vårdcentral, Huskvarna
  - Gränna vårdcentral, Jönköping
  - Lokstallarna vårdcentral, Jönköping
  - Norrahammars vårdcentral, Jönköping
  - Råslätts vårdcentral, Jönköping
  - Wetterhälsan, Jönköping
  - Kvarnholmens hälsocentral, Kalmar
  - Kärna vårdcentral, Linköping
  - Linghems vårdcentral, Linköping
  - Tannefors vårdcentral, Linköping
  - Stora Trädgårdsgatans hälsocentral, Västervik
  - Aroma Vårdcentral, Vetlanda

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon request to the principal investigator (Andreas Stomby) if it is in accordance with Swedish and international law. Thus, all requests will be judged before IPD is eventually shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after the research group has conducted the planned analyses. Preliminary in year 2027.
Access Criteria: See above